CLINICAL TRIAL: NCT05091346
Title: An Open-Label, Multicenter, Phase 1b/2 Study of E7386 in Combination With Pembrolizumab in Previously Treated Subjects With Selected Solid Tumors
Brief Title: A Study of E7386 in Combination With Pembrolizumab in Previously Treated Participants With Selected Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7386-G000-201; 2021-001568-10 (EudraCT Number); MK-3475-C83 (Other: Merck Sharp & Dohme); 2023-505425-14 (Registry Identifier: CTIS)
Record Dates: First submitted 2021-10-14; First posted 2021-10-25 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2024-10

CONDITIONS: Melanoma; Carcinoma, Hepatocellular; Colorectal Neoplasms
Keywords: metastatic or unresectable melanoma; metastatic or unresectable hepatocellular carcinoma; metastatic or unresectable colorectal cancer; Solid tumors; E7386
MeSH Terms: conditions — Melanoma; Carcinoma, Hepatocellular; Colorectal Neoplasms; Neoplasm Metastasis | interventions — E-7386; pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b and 2: E7386 + Pembrolizumab (Experimental): Participants will receive E7386 twice daily (BID) along with pembrolizumab 200 mg intravenous (IV) infusion once every 3 weeks (Q3W) in 21-day treatment cycle until RP2D is determined in Phase 1b. The recommended dose for Phase 2 part of the study will be based on Phase 1b result. Participants will continue to receive study treatment in Phase 2 part until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the study.
  Interventions: Drug: E7386; Drug: Pembrolizumab
- Phase 2: E7386 + Pembrolizumab + Lenvatinib (Experimental): Participants will be randomized to receive E7386 Dose 1 (Cohort 1) or Dose 2 (Cohort 2) tablet, BID, orally in combination with pembrolizumab 200 mg Q3W IV infusion plus lenvatinib 8 mg capsule, orally, once daily (QD) continuously in 21-days treatment cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the study. The dose of treatment depends on tolerability data of both Cohorts.
  Interventions: Drug: E7386; Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: E7386 — E7386 tablet.
Drug: Pembrolizumab — Pembrolizumab IV infusion.
  Other Names: KEYTRUDA®
Drug: Lenvatinib — Lenvatinib capsule.
  Other Names: E7080
  Arms: Phase 2: E7386 + Pembrolizumab + Lenvatinib

SUMMARY:
The Phase 1b part of this study is conducted to assess the safety and tolerability of E7386 in combination with pembrolizumab in participants with previously treated selected solid tumors, and to determine the recommended Phase 2 dose (RP2D) of E7386 in combination with pembrolizumab.

The Phase 2 part of this study is conducted to assess the objective response rate (ORR) of E7386 in combination with pembrolizumab (melanoma, colorectal cancer [CRC], hepatocellular carcinoma [HCC]) or of E7386 in combination with pembrolizumab plus lenvatinib (HCC) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

ELIGIBILITY:
Inclusion Criteria

1. Male or female, age >=18 years at the time of informed consent
2. Have a histologically or cytologically-documented, advanced (metastatic and/or unresectable) selected solid tumor for which prior standard systemic therapy has failed. Selected tumor types: melanoma (excluding uveal melanoma), CRC, HCC
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Must have disease progression on current or since the last anticancer treatment
5. At least one measurable lesion by computer tomography (CT) or magnetic imaging resonance (MRI) based on RECIST 1.1
6. Adequate organ function and serum mineral level per blood work as confirmed by the investigator

   1. Calcium (albumin-corrected) within normal range
   2. Potassium within normal reference range
   3. Magnesium less than or equal to (>=) 1.2 milligram per deciliter (mg/dL) or 0.5 millimoles per litre (mmol/L).
7. Melanoma cohort (Phase 2), participants must have:

   * Unresectable Stage III or Stage IV melanoma, not amenable to local therapy.
   * Received only 1 or, if BRAF mut +ve, 2 lines of therapies locally advanced or metastatic setting prior to study enrolment. Note: Adjuvant anti-PD-1/PD-L1 mAb/ BRAF inhibitor treatment will be counted as prior line of treatment if relapse occurred during active treatment or within 12 weeks of treatment discontinuation.
8. CRC cohort (Phase 2), participants must have received at least 2 prior systemic therapies in adjuvant and/or metastatic setting (not exceeding 4 lines of therapies in the metastatic setting, progressed on at least 1 prior regimen in the metastatic setting or could not tolerate standard treatment)
9. Participants with HCC cohort (Phase 2) must have:

   * Stage B (not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment) or stage C based on Barcelona Clinic Liver Cancer [BCLC] staging System and Child-Pugh class A only.
   * Have received only 1 prior line of systemic therapy in the locally advanced or metastatic setting, and must have progressed on treatment with an anti-PD-1/L1 monoclonal antibodies (mAb) administered either as monotherapy, or in combination
10. Must agree to take Vitamin D continuous supplementation as per local institutional guideline/ investigator's clinical discretion if their 25-hydroxyvitamin D levels are less than 10 nanogram per milliliter (ng/mL).
11. Triplet treatment cohorts only: Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP <=150/90 millimeter of mercury (mmHg) at Screening/Baseline and no change in antihypertensive medications within 1 week before starting treatment in this study.

Exclusion Criteria

1. Have present or progressive accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to study drug administration. The participant can receive diuretic drugs as needed per the treating physician. Consult with the sponsor if the participant has more than trivial/trace fluid accumulation.
2. Prior treatment with E7386 or prior therapy with anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (example, CTLA-4, OX 40, CD137) that was discontinued due to a Grade 3 or higher immune-related (ir)AE
3. Participants with central nervous system (CNS) metastases are not eligible unless they are previously treated are radiologically stable, that is, without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), and are clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
4. Any active infection requiring systemic treatment
5. Have severe hypersensitivity to study drugs and/or any of its excipients
6. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Have an active autoimmune disease that has required systemic treatment in the past 2 years
8. Have a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
9. Any bone disease/conditions as follows:

   * Osteoporosis with T-score <-2.5 by DXA scan
   * Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia
   * Symptomatic hypercalcemia requiring bisphosphonate therapy
   * History of any fracture within 6 months prior to starting study drug
   * History of symptomatic vertebral fragility fracture or any fragility fracture
   * Moderate or severe morphometric vertebral fracture at baseline.
   * Any condition requiring orthopedic intervention.
   * Bone metastases not being treated with a bisphosphonate or denosumab
10. Active viral hepatitis (B or C) as demonstrated by positive serology for participants with melanoma and CRC. Dual active hepatitis B virus (HBV) infection and hepatitis C virus (HCV) infection at study entry for participants with HCC
11. Known to be human immunodeficiency virus (HIV) positive
12. Received blood/platelet transfusion or G-CSF within 4 weeks before study entry
13. For Melanoma only, participants with ocular melanoma are excluded. Note: Participants with mucosal melanoma will not exceed 20% of the enrolled participants in melanoma cohort in Phase 2.
14. For CRC only, participants are excluded if:

    - have a tumor that is microsatellite instability high (MSI H)/ DNA mismatch repair-deficient (dMMR) positive
15. For HCC only, participants are excluded if:

    * Clear invasion to bile duct
    * Have had esophageal or gastric variceal bleeding within the last 6 months. Participants in triplet treatment cohorts will be screened for esophageal or gastric varices unless such screening has been performed in the past 3 months before first dose of treatment. If varices are present, they should be treated according to institutional standards before starting study intervention; esophageal or gastric varices that require interventional treatment within 28 days prior to first dose of study drug are excluded
    * History of hepatic encephalopathy within 6 months prior to starting study drug unresponsive to therapy within 3 days. Participants on rifaximin or lactulose during screening to control their hepatic encephalopathy are not allowed
16. For participants in the triplet treatment cohorts only:

    * Proteinuria greater than (>) 1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein >=1 gram per 24 hours (g/24 hours) will be ineligible
    * Bleeding or thrombotic disorders or use of anticoagulants requiring therapeutic INR monitoring (example, warfarin or similar agents). Treatment with low molecular weight heparin and factor X inhibitors is permitted
    * Clinically significant hemoptysis from any source or tumor bleeding within 3 weeks prior to the first dose of study drug
    * Pre-existing >=Grade 3 gastrointestinal or non-gastrointestinal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (10):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine Health, Orange, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - SCRI Florida Cancer Specialists East, West Palm Beach, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Rutgers cancer Institute of NJ, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Providence Medical Center Institute Franz Clinic, Portland, Oregon
  - Tennessee Oncology PPLC, Nashville, Tennessee
- Japan (9):
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital, Chūōku
  - Kurume University Hospital, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - Osaka Metropolitan University Hospital, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Sapporo-Kosei General Hospital, Sapporo
  - Shizuoka Cancer Center Hospital, Shizouka
  - Toranomon Hospital, Tokyo
- Spain (9):
  - Hospital Regional Universitario de Malaga, Málaga, Avenida Carolos Haya S/n
  - Hospital Clínico San Carlos, Madrid, Calle Profesor Martín Lagos
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario de la Paz, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Imperial College London - Hammersmith Hospital, London
  - Royal Free Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in Japan, United States, Spain, and United Kingdom from 27 October 2021 to 15 October 2024.
Pre-assignment Details: A total of 152 participants were screened, of which 63 were screen failures and 89 received study treatment.
Groups:
- Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg: Participants received E7386 100 milligrams (mg), tablets, orally, twice daily (BID), plus pembrolizumab 200 mg, intravenous (IV) infusion, every 3 weeks (Q3W) continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg: Participants received E7386 120 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg: Participants with hepatocellular carcinoma (HCC) received E7386 120 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg: Participants with melanoma received E7386 120 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg: Participants with colorectal cancer (CRC) received E7386 120 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
Period: Overall Study
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
Started | 6 | 6 | 17 | 29 | 31
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 17 | 29 | 31
Not completed — Survival follow-up ceased/discontinued by sponsor | 0 | 0 | 7 | 10 | 4
Not completed — Death | 6 | 5 | 8 | 16 | 26
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Efficacy Analysis Set included all participants with measurable disease at Baseline who received at least 1 dose of any study drug.
Groups:
- Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg: Participants received E7386 100 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg: Participants with HCC received E7386 120 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg: Participants with CRC received E7386 120 mg, tablets, orally, BID, plus pembrolizumab 200 mg, IV infusion, Q3W continuously in 21-day cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice, or discontinuation of the study program.
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 6 | 6 | 17 | 29 | 31 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.38) | 63.3 (14.00) | 66.4 (12.52) | 60.8 (11.16) | 55.5 (11.20) | 60.5 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 10 | 12 | 35
  Male | 2 | 3 | 11 | 19 | 19 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 6 | 6 | 16 | 27 | 29 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 5 | 5 | 12 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 4 | 6
  White | 0 | 0 | 10 | 23 | 14 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b Part: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 based on investigator assessment. DLT was defined as any of the hematological or non-hematological toxicities events that: - Failure to administer greater than or equal to (>=) 75 percentage (%) of the planned dosage of E7386 as a result of treatment-related toxicity; - Any treatment-related toxicity that causes the participant to discontinue treatment, even if the toxicity does not meet DLT criteria; - Prolonged delay (greater than [>] 2 weeks) in initiating Cycle 2 due to treatment-related toxicities; - Any Grade 5 event or any death not clearly due to the underlying disease or extraneous causes.
Time Frame: Cycle 1 (Cycle length=21 days)
Population: The DLT Analysis Set included all participants in Phase 1b part who had received study drug as planned (that is [i.e.], complete at least 75% of the planned E7386) in Cycle 1, or who experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Primary Outcome: Phase 1b Part: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that emerged during treatment, having been absent at pretreatment (Baseline) or reemerged during treatment, or up to 30 days following last dose of study drug, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment or up to 30 days following last dose of study drug, relative to the pretreatment state, when the AE was continuous.
Time Frame: Up to 30 days after last dose of study drug (up to 12.73 months)
Population: Safety Analysis Set included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

3. Primary Outcome: Phase 1b Part: Number of Participants With Serious TEAEs
Description: An SAE was any untoward medical occurrence that at any dose: Resulted in death; Was life-threatening (i.e., the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death); Required inpatient hospitalization or prolongation of existing hospitalization; Resulted in persistent or significant disability/incapacity; Was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). An SAE was also counted as a TEAE if it emerged up to 90 days after the participant's last dose of study drug, or up to 30 days following cessation of study drug if the participant initiated new anticancer therapy, whichever was earlier.
Time Frame: Up to 90 days after last dose of study drug (up to 14.73 months)
Population: Safety Analysis Set included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 2

4. Primary Outcome: Phase 2 Part: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal (i.e., decrease in short axis to less than [<] 10 millimeters [mm]). PR: At least a 30 percent (%) decrease in sum of the diameters (SOD) of target lesions, taking as reference the screening SOD. Additionally, progression of target lesions must not be present.
Time Frame: Up to 20.40 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 17 | 29 | 31
percentage of participants | 0.0 [0.0 to 19.5] | 6.9 [0.8 to 22.8] | 3.2 [0.1 to 16.7]

5. Secondary Outcome: Phase 1b Part: Percentage of Participants With Best Overall Response (BOR)
Description: BOR was defined as CR, PR, stable disease (SD), progressive disease (PD), and not applicable (NA)/not evaluable (NE) as per RECIST version 1.1. CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal (i.e., decrease in short axis to <10 mm). PR: At least a 30% decrease in SOD of target lesions, taking as reference screening SOD. Additionally, progression of target lesions must not be present. SD: Neither sufficient shrinkage of target lesions to qualify for PR, nor sufficient increase to qualify for PD. PD: At least a 20% increase in the SOD of target lesions, taking as reference nadir SOD (or the screening, if screening is nadir value). In addition to relative increase of 20% in SOD, the SOD must also demonstrate an absolute increase of >=5 mm. NA: No target lesions were identified at Screening.
Time Frame: Up to 11.73 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
percentage of participants
  CR | 0 | 0
  PR | 0 | 0
  SD | 83.3 | 33.3
  PD | 16.7 | 50.0
  NA/NE | 0 | 16.7

6. Secondary Outcome: Phase 1b and Phase 2 Parts: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of CR or PR to the first documentation of PD or death due to any cause (whichever occurs first), in participants with confirmed CR or PR per RECIST 1.1. CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal (i.e., decrease in short axis to <10 mm). PR: At least a 30% decrease in SOD of target lesions, taking as reference screening SOD. Additionally, progression of target lesions must not be present. SD: Neither sufficient shrinkage of target lesions to qualify for PR, nor sufficient increase to qualify for PD. PD: At least a 20% increase in the SOD of target lesions, taking as reference nadir SOD (or the screening, if screening is nadir value). In addition to relative increase of 20% in SOD, the SOD must also demonstrate an absolute increase of >=5 mm.
Time Frame: Phase 1b Part: Up to 11.73 months; Phase 2 Part: Up to 20.40 months
Population: Efficacy Analysis Set included all participants with measurable disease at Baseline who received at least 1 dose of any study drug. Here, "Overall Number of Participants Analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1
months |  |  |  | 14.1 [12.4 to NA] — Here, "NA" means upper limit of confidence interval could not be estimated due to low number participants with events. | 7.5 [NA to NA] — Here, "NA" means upper and lower limit of confidence interval could not be estimated due to low number participants with events.

7. Secondary Outcome: Phase 1b and Phase 2 Parts: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had a best overall response of confirmed CR or PR, or SD (after >=5 weeks from the first dose) as per RECIST 1.1. CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal (i.e., decrease in short axis to <10 mm). PR: At least a 30% decrease in SOD of target lesions, taking as reference screening SOD. Additionally, progression of target lesions must not be present. SD: Neither sufficient shrinkage of target lesions to qualify for PR, nor sufficient increase to qualify for PD. PD: At least a 20% increase in the SOD of target lesions, taking as reference nadir SOD (or the screening, if screening is nadir value). In addition to relative increase of 20% in SOD, the SOD must also demonstrate an absolute increase of >=5 mm.
Time Frame: Phase 1b Part: Up to 11.73 months; Phase 2 Part: Up to 20.40 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6 | 17 | 29 | 31
percentage of participants | 83.3 [35.9 to 99.6] | 33.3 [4.3 to 77.7] | 58.8 [32.9 to 81.6] | 48.3 [29.4 to 67.5] | 32.3 [16.7 to 51.4]

8. Secondary Outcome: Phase 1b and Phase 2 Parts: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants who had a best overall response of confirmed CR or PR, or durable SD (duration of SD >=23 weeks) per RECIST 1.1. CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal (i.e., decrease in short axis to <10 mm). PR: At least a 30% decrease in SOD of target lesions, taking as reference screening SOD. Additionally, progression of target lesions must not be present. SD: Neither sufficient shrinkage of target lesions to qualify for PR, nor sufficient increase to qualify for PD.
Time Frame: Phase 1b Part: Up to 11.73 months; Phase 2 Part: Up to 20.40 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6 | 17 | 29 | 31
percentage of participants | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 11.8 [1.5 to 36.4] | 13.8 [3.9 to 31.7] | 16.1 [5.5 to 33.7]

9. Secondary Outcome: Phase 2 Part: Number of Participants With TEAEs and Treatment-related TEAEs
Description: A TEAE was defined as an AE that emerged during treatment, having been absent at pretreatment (Baseline) or reemerged during treatment, or up to 30 days following last dose of study drug, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment or up to 30 days following last dose of study drug, relative to the pretreatment state, when the AE was continuous. Related TEAEs was defined as AE for which a causal relationship between the study drug and the AE was a reasonable possibility.
Time Frame: Up to 30 days after last dose of study drug (up to 21.40 months)
Population: Safety Analysis Set included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 17 | 29 | 31
Participants
  TEAEs | 17 | 28 | 30
  Treatment Related TEAEs | 16 | 26 | 28

10. Secondary Outcome: Phase 1b Part, Cmax: Maximum Observed Plasma Concentration for E7386 When Co-administered With Pembrolizumab
Description: Cmax was defined as the maximum plasma concentration for E7386 when co-administered with Pembrolizumab. PK parameters were derived by noncompartmental analysis.
Time Frame: Cycle 1 Days 1 and 8: Pre-dose up to 12 hours post-dose (Cycle 1 length=21 days)
Population: Pharmacokinetic Analysis Set included all participants who had received at least 1 dose of study drug and had at least 1 evaluable plasma E7386 concentration. As planned, this PK parameter was assessed in Phase 1b Part only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 401 (232.0) | 472 (82.1)
  Cycle 1 Day 8 | 386 (240.0) | 706 (86.4)

11. Secondary Outcome: Phase 1b Part, Tmax: Time to Reach the Maximum Plasma Concentration for E7386 When Co-administered With Pembrolizumab
Description: Tmax was defined as the time to reach maximum observed plasma concentration for E7386 when co-administered with Pembrolizumab. PK parameters were derived by noncompartmental analysis.
Time Frame: Cycle 1 Days 1 and 8: Pre-dose up to 12 hours post-dose (Cycle 1 length=21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
hour
  Cycle 1 Day 1 | 0.70 [0.35 to 5.93] | 2.00 [0.53 to 2.05]
  Cycle 1 Day 8 | 2.90 [1.90 to 3.93] | 1.38 [0.55 to 6.00]

12. Secondary Outcome: Phase 1b Part, AUC(0-t): Area Under the Plasma Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for E7386 When Co-administered With Pembrolizumab
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from 0 (pre-dose) to time of last quantifiable concentration for E7386 when co-administered with Pembrolizumab. PK parameters were derived by noncompartmental analysis.
Time Frame: Cycle 1 Days 1 and 8: Pre-dose up to 12 hours post-dose (Cycle 1 length=21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
nanogram*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 874 (192.0) | 1400 (52.5)
  Cycle 1 Day 8 | 1830 (180.0) | 2540 (81.3)

13. Secondary Outcome: Phase 1b Part, CLss/F: Apparent Clearance From Plasma at Steady State for E7386 When Co-administered With Pembrolizumab
Description: CLss/F for E7386 when co-administered with Pembrolizumab was reported. PK parameters were derived by noncompartmental analysis.
Time Frame: Cycle 1 Day 8: Pre-dose up to 12 hours post-dose (Cycle 1 length=21 days)
Population: Pharmacokinetic Analysis Set included all participants who had received at least 1 dose of study drug and had at least 1 evaluable plasma E7386 concentration. As planned, this PK parameter was assessed in Phase 1b Part at Cycle 1 Day 8 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 6
liter per hour | 54.0 (181.0) | 46.9 (80.7)

ADVERSE EVENTS:
Time Frame: Non-serious: Up to 30 days after last dose of the study drug (up to 12.73 months for Phase 1b and up to 21.40 months for Phase 2); All-cause Mortality and SAEs: Up to 90 days after last dose of the study drug (up to 14.73 months for Phase 1b and 23.40 months for Phase 2)
Arm/Group | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/6 | 8/17 | 16/29 | 26/31
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 7/17 | 5/29 | 10/31
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 17/17 | 28/29 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg (N=6) | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg (N=6) | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg (N=17) | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg (N=29) | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg (N=31)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Liver function test abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b, Dose Escalation: E7386 100 mg + Pembrolizumab 200 mg (N=6) | Phase 1b, Dose Escalation: E7386 120 mg + Pembrolizumab 200 mg (N=6) | Phase 2, Dose Expansion, HCC: E7386 120 mg + Pembrolizumab 200 mg (N=17) | Phase 2, Dose Expansion, Melanoma: E7386 120 mg + Pembrolizumab 200 mg (N=29) | Phase 2, Dose Expansion, CRC: E7386 120 mg + Pembrolizumab 200 mg (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 5 (8) | 6 (20) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6) | 5 (5) | 3 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 7 (12) | 10 (14) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 8 (10) | 9 (17) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (8) | 4 (5) | 15 (30) | 18 (35) | 19 (27)
Vomiting (Gastrointestinal disorders) | 4 (11) | 5 (7) | 12 (30) | 22 (49) | 18 (36)
Asthenia (General disorders) | 0 (0) | 0 (0) | 4 (7) | 10 (16) | 3 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 7 (17)
Malaise (General disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (4)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (3) | 1 (2) | 0 (0) | 2 (4) | 6 (9)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 4 (6) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 5 (7) | 4 (4) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (7)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (10)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 3 (7) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 5 (7) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 3 (3) | 7 (14) | 10 (12)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 6 (13) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT05091346/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT05091346/SAP_001.pdf